CLINICAL TRIAL: NCT04069819
Title: Double-blind, Randomized, Placebo-Controlled Pilot Study of the Phosphodiesterase-3 Inhibitor Cilostazol as an Adjunctive to Antidepressants in Patients With Major Depressive Disorder
Brief Title: The Phosphodiesterase-3 Inhibitor Cilostazol as an Adjunctive to Antidepressants in Patients With Major Depressive Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUR22021
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cilostazol; Tablets; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Escitalopram 20 mg tablet once daily for 6 week plus placebo tablet twice daily for 6 weeks
  Interventions: Drug: Escitalopram; Drug: Placebo
- Cilostazol group (Experimental): Escitalopram 20 mg tablet once daily for 6 week plus Cilostazol 50mg tablet twice daily for 6 weeks
  Interventions: Drug: Cilostazol 50 MG Oral Tablet; Drug: Escitalopram

INTERVENTIONS:
Drug: Cilostazol 50 MG Oral Tablet — Escitalopram,Selective serotonin reuptake inhibitor- Cilostazol, a selective phosphodiesterase 3 (PDE3) inhibitor, acts as an antiplatelet agent and has been widely approved for treatment of intermittent claudication with peripheral arterial disease and for secondary prevention of ischemic stroke.
  Arms: Cilostazol group
Drug: Escitalopram — Escitalopram 20 mg tablet once daily for 6 week
Drug: Placebo — placebo
  Arms: Control group

SUMMARY:
Cilostazol is a PDE 3 inhibitor, which showed as decrease in HAM-D scores in post-stroke depression through inhibition of neurodegeneration in the primary lesion and secondary extrafocal sites and through promotion of neurogenesis. These beneficial effects on post-stroke depression may be involved in activation of CREB/BDNF signaling.The aim of the current study is to evaluate the potential adjunct antidepressant effect of cilostazol in adult patients with MDD. Furthermore, we will assess the relationship between HAM-D score and BDNF as well as their role as a therapeutic targets of MDD.

DETAILED DESCRIPTION:
Cilostazol produces various powerful pleiotropic effects via restoration of intracellular second messenger cyclic adenosine monophosphate (cAMP). Treatment with cilostazol against cerebral ischemic injury ameliorates negative effects of cerebral hypoperfusion through the PDE3- cAMP signaling cascade with subsequent activation of inducible transcription factor cAMP response element-binding protein (CREB), suggesting the importance of the CREB signaling pathway.

Activation of CREB promotes the gene expression of neuroprotective molecules that activate subsequent anti-apoptotic pathways with the gene expression of brain-derived neurotrophic factor (BDNF). BDNF also regulates neurogenesis, proliferation, and survival of neural stem or progenitor cells, as well as neuronal survival. In addition, CREB and BDNF signaling play an important role in the pathophysiology of major depressive disorder .

Psychopharmacotherapy with antidepressants or mood stabilizers provides an effective treatment for depression after stroke, but alternative therapy by activation of CREB and BDNF signaling may exert beneficial effects on various aspects of negative mood. Drugs that activate CREB and BDNF signaling may provide a potential therapeutic approach for treatment of poststroke depression via neural cell survival and proliferation of neural progenitor cells.

The aim of the current study is to evaluate the potential adjunct antidepressant effect of cilostazol in adult patients with MDD. Furthermore, we will assess the relationship between HAM-D score and BDNF as well as their role as a therapeutic targets of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 20 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).
* Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females
* Cardiovascular disorders
* Severe renal impairment: creatinine clearance of ≤ 25 ml/min
* Moderate or severe hepatic impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 6 weekS
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
Effect on biological markers | 6 week
  Serum level of brain derived neurotrophic factor (BDNF), cAMP response element-binding protein (CREB), SEROTONIN, tumor necrosis factor alpha (TNF-α), Interleukin-6 (IL-6), and Nuclear factor kappa were measured at the baseline and after the treatment to evaluate the biological effects of the used medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Abdallah MS, Ramadan AN, Omara-Reda H, Mansour NO, Elsokary MA, Elsawah HK, Zaki SA, Abo Mansour HE, Mosalam EM. Double-blind, randomized, placebo-controlled pilot study of the phosphodiesterase-3 inhibitor cilostazol as an adjunctive to antidepressants in patients with major depressive disorder. CNS Neurosci Ther. 2021 Dec;27(12):1540-1548. doi: 10.1111/cns.13731. Epub 2021 Sep 21. PMID 34545997